CLINICAL TRIAL: NCT06761560
Title: Optimizing Hydroxyurea Dosage With Pharmakokinetic in Patients Suffering of Moderate to Severe Sickle Cell Anemia
Acronym: OPTIMA
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yves Pastore (Other)
Collaborators: St. Justine's Hospital (Other)
Responsible Party: Sponsor-Investigator, Yves Pastore, Co-director Sickle Cell Programm, Principal Investigator, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-4674
Record Dates: First submitted 2024-12-12; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Sickle Cell Disease (SCD)
Keywords: hydroxyurea; pharmacokinetic; sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Group A will receive dosing of hydroxyurea depending on the HU-AUC result at different timepoint until MTD Group B will receive dosing of hydroxyurea following the standard of care bloodwork follow-up until MTD Group C will undergo one pharmacokinetic testing after taking hydroxyurea for at least 12 months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Patient starting hydroxyurea that will have PK sample procurements at different timpoints over a period of 12 months until HU-AUC shows MTD
  Interventions: Diagnostic Test: Pharmacokinetic based dosage change
- Group B (No Intervention): Patient starting hydroxuyrea that will be followed as per standard of care over a period of 12 months until MTD has been reached
- Group C (Experimental): Patient will undergo one PK sample procurement to evaluate level of HU-AUC after 12 months of taking hydroxyurea.
  Interventions: Diagnostic Test: Pharmacokinetic dosing

INTERVENTIONS:
Diagnostic Test: Pharmacokinetic based dosage change — This study will compare 2 groups of sickle cell patients that are receiving hydroxyurea. Group A will have an increase in their dosage based on the pharmacokinetic result over a period of 12 months and Group B will have an increase in their dosage based on the standard of care follow-up over a period of 12 months. The aim is to evaluate if the group A can reach MTD faster than than the Group B
  Arms: Group A
Diagnostic Test: Pharmacokinetic dosing — Patient with sickle cell disease will undergo one pharmacokinetic test after taking 12 months of hydroxyurea to evaluate HU-AUC at that timepoint
  Arms: Group C

SUMMARY:
The goal of this study is to evaluate if patients with sickle cell disease can achieve a maximum tolerate dose of hydroxuyrea (HU) over a period of 12 months faster with pharmacokinetic testing than the standard of care bloodwork follow-up. Pharmacokinetic test is used to evaluate the process by which drugs are absorbed, distributed in the body, localized in the tissues, and is excreted.

Patient will be a randomized (coin toss method) into 2 groups. Group A will have an increase of their HU dosage with pharmacokinetic results and Group B will have an increase of their HU dosage following the standard of care bloodwork follow-up.

Group C will include patient with sickle cell disease that has been taking HU for at least 12 months and will undergo a pharmacokinetic dosage to check the level of HU only one time.

ELIGIBILITY:
Inclusion Criteria (Group A and B) :

* Have had confirmed diagnosis of SCD at CHU Sainte-Justine biochemistry lab with hemoglobin electrophoresis.
* Be patients with SS, SBThal0.
* Agree to take hydroxyurea for a period of 12 months
* Be between age of 6months old and 18 years old.
* Have consented for participation in the study.

Inclusion Criteria (Group C) :

* Have had confirmed diagnosis of SCD at CHU Sainte-Justine biochemistry lab with hemoglobin electrophoresis.
* Be patients with SS, SBThal0.
* Have taken hydroxyurea for a period of at least 12 months, and have received HU at a stable dose and at MTD for at least 6 months.
* Be between age of 6months old and 18 years old.
* Have consented for participation in the study.

Exclusion Criteria:

* Patients with sickle cell genotype other than SS or SBThal0 (SC, SBThal+, SE or SD)
* Patients on chronic transfusion program
* Patients have received a blood transfusion in the last 4 weeks of study enrollment.
* Have received a hematopoietic stem-cell transplantation
* Creatinine >2x normal for age
* ALT>2x normal for age
* Sexually active females unwilling to comply with reliable method of birth control
* Pregnancy
* Conditions which in the opinion of the investigator, would compromise participation in the study will be excluded.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2027-11-25 (Estimated); Study Completion 2027-11-25 (Estimated)

PRIMARY OUTCOMES:
Evaluation of HU-PK at 6 months between group A and group B | At 6 months
  Pharmakocinetic dosage of hydroxyurea will be determined at 6 months in group A and group B. We hypothesize that HU-PK in group B may be lower (suboptimal) compared to group A.

SECONDARY OUTCOMES:
Time to reach maximal tolerated dose (MTD) | 3, 6, 9 and 12 months
  Time (weeks) to achieve MTD in groups A and B will be determined by evaluating the % of patients reaching MTD (at 3 , 6, 9 and 12 months) in each group.
  MTD is defined by hematological parameters: Absolute neutrophile count 0.8-1.5x10*9/L or platelet 80-120x10*9/L or absolute reticulocyte count 50-80x10*9/L)
Fetal hemoglobin | at 3, 6 and 12 months
  Comparing fetal hemoglobin between group A and B
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) in group A and B | From enrollment to 12 months
  Evaluation of the incidence adverse events (AE) and serious adverse events (SAE) in both groups
Evaluation of % of patients reaching AUC of 115 +/- 15mg*h/L at 12 months compared to the percentage of patients in group C reaching the same AUC | At 12 months
  Percentage of patients in the HU-AUC (group A) with an AUC of 115 mg*h/L at 12 months will be compared to the percentage of patients in group C with an AUC of 115 +/-15 mg*h/L.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
This is a pilot study with a small group of participant.

REFERENCES:
- [Background] Verduzco LA, Nathan DG. Sickle cell disease and stroke. Blood. 2009 Dec 10;114(25):5117-25. doi: 10.1182/blood-2009-05-220921. PMID 19797523
- [Background] Meier ER. Treatment Options for Sickle Cell Disease. Pediatr Clin North Am. 2018 Jun;65(3):427-443. doi: 10.1016/j.pcl.2018.01.005. PMID 29803275
- [Background] McGann PT, Niss O, Dong M, Marahatta A, Howard TA, Mizuno T, Lane A, Kalfa TA, Malik P, Quinn CT, Ware RE, Vinks AA. Robust clinical and laboratory response to hydroxyurea using pharmacokinetically guided dosing for young children with sickle cell anemia. Am J Hematol. 2019 Aug;94(8):871-879. doi: 10.1002/ajh.25510. Epub 2019 Jun 12. PMID 31106898
- [Background] Dong M, McGann PT. Changing the Clinical Paradigm of Hydroxyurea Treatment for Sickle Cell Anemia Through Precision Medicine. Clin Pharmacol Ther. 2021 Jan;109(1):73-81. doi: 10.1002/cpt.2028. Epub 2020 Oct 8. PMID 32869281
- [Background] Marahatta A, Ware RE. Hydroxyurea: Analytical techniques and quantitative analysis. Blood Cells Mol Dis. 2017 Sep;67:135-142. doi: 10.1016/j.bcmd.2017.08.009. Epub 2017 Aug 8. PMID 28847416
- [Background] Hai X, Guo M, Gao C, Zhou J. Quantification of hydroxyurea in human plasma by HPLC-MS/MS and its application to pharmacokinetics in patients with chronic myeloid leukaemia. J Pharm Biomed Anal. 2017 Apr 15;137:213-219. doi: 10.1016/j.jpba.2017.01.008. Epub 2017 Jan 10. PMID 28131939
- [Background] Wang WC, Ware RE, Miller ST, Iyer RV, Casella JF, Minniti CP, Rana S, Thornburg CD, Rogers ZR, Kalpatthi RV, Barredo JC, Brown RC, Sarnaik SA, Howard TH, Wynn LW, Kutlar A, Armstrong FD, Files BA, Goldsmith JC, Waclawiw MA, Huang X, Thompson BW; BABY HUG investigators. Hydroxycarbamide in very young children with sickle-cell anaemia: a multicentre, randomised, controlled trial (BABY HUG). Lancet. 2011 May 14;377(9778):1663-72. doi: 10.1016/S0140-6736(11)60355-3. PMID 21571150
- [Background] Thornburg CD, Files BA, Luo Z, Miller ST, Kalpatthi R, Iyer R, Seaman P, Lebensburger J, Alvarez O, Thompson B, Ware RE, Wang WC; BABY HUG Investigators. Impact of hydroxyurea on clinical events in the BABY HUG trial. Blood. 2012 Nov 22;120(22):4304-10; quiz 4448. doi: 10.1182/blood-2012-03-419879. Epub 2012 Aug 22. PMID 22915643
- [Background] Yahouedehou SCMA, Adorno EV, da Guarda CC, Ndidi US, Carvalho SP, Santiago RP, Aleluia MM, de Oliveira RM, Goncalves MS. Hydroxyurea in the management of sickle cell disease: pharmacogenomics and enzymatic metabolism. Pharmacogenomics J. 2018 Dec;18(6):730-739. doi: 10.1038/s41397-018-0045-1. Epub 2018 Sep 12. PMID 30206297
- [Background] Switzer JA, Hess DC, Nichols FT, Adams RJ. Pathophysiology and treatment of stroke in sickle-cell disease: present and future. Lancet Neurol. 2006 Jun;5(6):501-12. doi: 10.1016/S1474-4422(06)70469-0. PMID 16713922
- [Background] Quinn CT. Sickle cell disease in childhood: from newborn screening through transition to adult medical care. Pediatr Clin North Am. 2013 Dec;60(6):1363-81. doi: 10.1016/j.pcl.2013.09.006. PMID 24237976
- [Background] Hebbel RP. Ischemia-reperfusion injury in sickle cell anemia: relationship to acute chest syndrome, endothelial dysfunction, arterial vasculopathy, and inflammatory pain. Hematol Oncol Clin North Am. 2014 Apr;28(2):181-98. doi: 10.1016/j.hoc.2013.11.005. PMID 24589261
- [Background] Kuypers FA. Hemoglobin s polymerization and red cell membrane changes. Hematol Oncol Clin North Am. 2014 Apr;28(2):155-79. doi: 10.1016/j.hoc.2013.12.002. Epub 2014 Jan 22. PMID 24589260
- [Background] Pleasants S. Epidemiology: a moving target. Nature. 2014 Nov 13;515(7526):S2-3. doi: 10.1038/515S2a. No abstract available. PMID 25390139
- See also: Related Info — https://www.chudequebec.ca/patient/maladies-soins-et-services/m-informer-sur-les-soins-et-services/programme-quebecois-de-depistage-neonatal-sanguin.aspx